CLINICAL TRIAL: NCT02470845
Title: A Randomized Controlled Trial of Tian Jiu Therapy for Allergic Rhinitis
Brief Title: Trial of Tian Jiu Therapy for Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Professor, Director of Clinical Division,, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJAR001
Record Dates: First submitted 2015-05-17; First posted 2015-06-12 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Allergic Rhinitis (AR)
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tian Jiu group (Experimental): The TJ group will undergo a 4-week treatment with herbal patches one session per week and a 4-week post-treatment follow-up, of one assessment session per week. Participants in the TJ group will be treated with herbal patches of Tian Jiu group on five acupoints on the back.
  Interventions: Drug: herbal patches of Tian Jiu group
- Placebo-control group (Sham Comparator): The placebo-control group will undergo a 4-week treatment with placebo patches one session per week and a 4-week post-treatment follow-up, of one assessment session per week. Participants in this group will be treated with placebo patches of placebo-control group on the same acupionts as the TJ group.
  Interventions: Drug: placebo patches of placebo-control group
- Waitlist-control group (No Intervention): The waitlist-control group will receive no treatment during the first 4 weeks but, beginning with the 5th week this group will receive TJ treatment for four weeks as compensatory.

INTERVENTIONS:
Drug: herbal patches of Tian Jiu group — The formula of herbal patch consists of BaiJieZi (Sinapis Semen), Yan Hu Suo（CorydulisRhizoma）、ZhiGan Sui (Kansui Radix)、Xi Xin (Asari Radix et rhizama) and Rengong She xiang(Moschus Artifactus) . The four herbs will be ground into powder, mixed thoroughlywith 20% BaiJieZi (Sinapis Semen), 25% Yan Hu Suo（CorydulisRhizoma), 15% ZhiGan Sui (Kansui Radix), and 40% Xi Xin (Asari Radix et rhizama), and the mixed powder will mix with fresh ginger juice in the ratio of 20g to 25 ml. The mixture will be made to a patch weighted as 2g and 1cm*1cm round size. 0.02g artificial She Xiang (Moschus Artifactus) will be added on top of each patch. Each patch will be applied on one acupoint.
  Arms: Tian Jiu group
Drug: placebo patches of placebo-control group — The placebo patch consists of flour and edible pigments. These two ingredients will be mixed with water and made to patches weighted as 2g and 1cm*1cm round size.Each patch will be applied on one acupoint.
  Arms: Placebo-control group

SUMMARY:
The aim of this study is to investigate the efficacy and safety of Tian Jiu in the treatment of allergic rhinitis compared with placebo and waitlist patients in Hong Kong.

DETAILED DESCRIPTION:
This will be a prospective, randomized, single-blinded, controlled trial in patients with AR. After a one-week run-in period, eligible subjects will be randomly assigned to the Tian Jiu group, placebo-control group and waitlist-control group. The TJ and placebo-control groups will undergo a 4-week treatment with one session per week and one 4-week post-treatment follow-up. Participants in the waitlist-control group will not receive any treatment during the first 4 weeks but will be required to be assessed. The total study period will be nine weeks.

ELIGIBILITY:
Inclusion Criteria:

* Positive skin prick tests
* High circulating levels of allergen-specific IgE antibody detected by a specific blood test for allergy called radioallergosorbent test (RAST)]
* Clinical history or allergen to have been identified
* Nasal provocation (test)

Exclusion Criteria:

* Allergic asthma, moderate to severe atopic dermatitis, autoimmune disorders, severe chronic inflammatory diseases, history of anaphylactic reactions, hypersensitivity to cetirizine or related drugs, specific immunotherapy during the past 3 years or planned in the next 2 years, pregnancy or breastfeeding.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change of total nasal symptom score | 4 weeks
  The change in the weekly average of total nasal symptom score (TNSS) recorded in participants' diaries from baseline（ Week 0） to end of the treatment（ Week 4）and post-treatment follow-up ( Week 8)

SECONDARY OUTCOMES:
Change of the Rhinitis Quality of Life Questionnaire (RQLQ) | 8 weeks
  The change in symptoms will be measured using the Rhinitis Quality of Life Questionnaire (RQLQ), by comparing the baseline( Week 0) with the scores within treatment (Week 2, 3), end of treatment( Week 4) and post-treatment follow-up ( Week 8).
Change in need for medication | 8 weeks
  The change in need for medication will be measured using an RM score (RMS), by comparing the baseline (Week 0) with the scores within treatment (Week 2, 3), end of treatment( Week 4) and post-treatment follow-up ( Week 8).

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Xiang Bian, Ph.D., M. D., Principal Investigator — School of Chinese Medicine, Hong Kong Baptist University
Locations (1):
- Hong Kong Baptist University Chinese Medicine Clinic, Hong Kong, China

REFERENCES:
- [Derived] Kun W, Zhong LL, Dai L, Cheng CW, Lu AP, Bian ZX. Tian Jiu therapy for allergic rhinitis: study protocol for a randomized controlled trial. Trials. 2016 May 17;17(1):248. doi: 10.1186/s13063-016-1374-5. PMID 27189087